CLINICAL TRIAL: NCT05150652
Title: Phase 2 Study of Neoadjuvant Endocrine Therapy in ER-positive, HER2-negative Early Stage Breast Cancer
Brief Title: Neoadjuvant Endocrine Therapy in ER-positive, HER2-negative Early Stage Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Irada Ibrahim-zada (Other)
Responsible Party: Sponsor-Investigator, Irada Ibrahim-zada, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21-BRE-54
Record Dates: First submitted 2021-11-24; First posted 2021-12-09 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; HER2-negative Breast Cancer; Node-negative Breast Cancer; Breast Carcinoma
Keywords: Neoadjuvant endocrine therapy; Early stage
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Letrozole; exemestane; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant Endocrine Therapy (Experimental): Participants will begin treatment with Anastrozole. If not tolerated well, participants will discontinue and begin treatment using Letrozole. If not tolerated well, participants will discontinue and begin treatment using Exemestane. If not tolerated well, participants will discontinue and begin treatment on Tamoxifen.
  Interventions: Drug: Anastrozole 1mg; Drug: Letrozole 2.5mg; Drug: Exemestane 25 mg; Drug: Tamoxifen

INTERVENTIONS:
Drug: Anastrozole 1mg — Participants will take 1mg of anastrozole once daily, orally, for up to six cycles of 28 days.
  Other Names: Arimidex
Drug: Letrozole 2.5mg — Participants will take 2.5mg of Letrozole once daily, orally, for up to six cycles of 28 days.
  Other Names: Femara
Drug: Exemestane 25 mg — Participants will take 25mg of Exemestane once daily, orally, for up to six cycles of 28 days.
  Other Names: Aromasin
Drug: Tamoxifen — Participants will take 20mg of Tamoxifen once daily, orally, for up to six cycles of 28 days.
  Other Names: Soltamox

SUMMARY:
The goal of this study is to access whether treatment of early state estrogen-rich breast cancers with neoadjuvant endocrine therapy will result in higher rates of margin negativity on lumpectomy specimen.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed invasive breast cancer, clinically stage I-II.
* Clinically lymph node negative
* Eligible for anti-endocrine treatment (per medical oncologist)
* Postmenopausal women
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Progesterone receptor negativity
* High grade tumor
* Synchronous non-breast malignancy
* Receiving any other investigational agents that could impact the efficacy of this trial regimen
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Anastrozole, Letrozole, Exemestane, Tamoxifen or other agents used in study
* Uncontrolled intercurrent illness
* Medical, psychiatric or other condition and/or social situations that would limit compliance with study requirements

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2026-06-09 (Estimated)

PRIMARY OUTCOMES:
Change in margin status | Baseline, 6-months after neoadjuvant treatment and surgery
  Evaluate the effect of neoadjuvant endocrine therapy (6-months course) on margin status of breast conservation surgery for women with early stage, low-risk breast cancer, defined as ER-positive, HER2-negative, node-negative breast carcinoma (single lesion only). Negative margin status is defined as no tumor on ink.

SECONDARY OUTCOMES:
Residual cancer burden | After neoadjuvant treatment and surgery (approximately 6 months from diagnosis)
  The following parameters are required from pathologic examination in order to calculate Residual Cancer Burden (RCB) after neoadjuvant treatment: Primary tumor bed area, overall cancer cellularity (as percentage of area), percentage of cancer that is in situ disease, number of positive lymph nodes and diameter of largest metastasis. These parameters are filled in in the calculator that is available online to calculate the Residual Cancer Burden index: http://www3.mdanderson.org/app/medcalc/index.cfm?pagename=jsconvert3
Pattern of response | After neoadjuvant treatment and surgery (approximately 6 months from diagnosis)
  Pattern of response (pathologic complete response, concentric shrinking with similar cellularity, size unchanged with decreased cellularity, no treatment response)
Change in satisfaction with cosmetic outcome | After neoadjuvant treatment and surgery (approximately 6 months and 12 months post-surgery)
  The Breast-Q© is a patient reported outcome measure for breast surgery that measures patient reported satisfaction and quality of life (QOL) developed by Memorial Sloan Kettering Cancer Center. It is comprised of 10 scales that address: 1) psychosocial well-being, 2) sexual well-being, 3) satisfaction with breasts, 4) physical well-being, 5) adverse effects of radiation, 6) satisfaction with information - breast surgeon, 7) satisfaction with information - radiation oncologist, 8) satisfaction with surgeon, 9) satisfaction with medical team, 10) satisfaction with office staff. Each module is scored from 0-100 where higher scores reflect a better outcome.

OTHER OUTCOMES:
Change in largest caliper measurement | Baseline, 6-months after neoadjuvant treatment and surgery
  Largest caliper measurement (millimeters) on post-therapy imaging vs. largest final size of tumor

CONTACTS AND LOCATIONS:
Overall Officials: Irada Ibrahim-zada, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDonald HG, Cassim EB, Harper MM, Burke EE, Marcinkowski EF, Cavnar MJ, Pandalai PK, Kim J. The Development of Investigator-Initiated Clinical Trials in Surgical Oncology. Surg Oncol Clin N Am. 2023 Jan;32(1):13-25. doi: 10.1016/j.soc.2022.07.003. Epub 2022 Nov 3. PMID 36410913